CLINICAL TRIAL: NCT04068844
Title: Mechanisms of Exercise Intolerance in Heart Failure With Preserved Ejection Fraction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: The University of Texas at Arlington (Other)
Responsible Party: Principal Investigator, Benjamin Levine, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: STU-2019-0617
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure, Diastolic
Keywords: Exercise; Hemodynamics,; Heart failure
MeSH Terms: conditions — Heart Failure, Diastolic; Motor Activity; Heart Failure | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: HFpEF patients with either central or peripheral limitations to exercise will be randomly assigned to either whole body or isolated single leg exercise.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Central HFpEF whole body exercise (Experimental): HFpEF patients who have a central limitation as the cause of the exercise intolerance randomized to whole body cycle training.
  Interventions: Behavioral: Exercise training
- Central HFpEF isolated single leg exercise (Experimental): HFpEF patients who have a central limitation as the cause of the exercise intolerance randomized to isolated single leg training.
  Interventions: Behavioral: Exercise training
- Peripheral HFpEF whole body exercise (Experimental): HFpEF patients who have a peripheral limitation as the cause of the exercise intolerance randomized to whole body cycle training.
  Interventions: Behavioral: Exercise training
- Peripheral HFpEF isolated single leg exercise (Experimental): HFpEF patients who have a peripheral limitation as the cause of the exercise intolerance randomized to isolated single leg training.
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training — Exercise training, either whole body or isolated single leg

SUMMARY:
The global objective of this study is to determine the mechanisms of exercise intolerance and dyspnea on exertion (DOE) in patients with HFpEF and based on this pathophysiology, test whether specific exercise training programs (whole body vs single leg) will result in improved exercise tolerance.

DETAILED DESCRIPTION:
This will be a randomized, non-blinded prospective intervention testing the effects of two types of exercise training, whole body and isolated single leg, on HFpEF patients with either central or peripheral limitations to exercise training. Subjects will undergo baseline maximal exercise testing and invasive right heart catheterization to define exercise tolerance and pulmonary and cardiac pressures during exercise. Based on the results of baseline testing, subjects will be divided into either centrally limited, defined as excessive rise in pulmonary capillary wedge pressure more than 25 mmHg that decreases after administration of sub-lingual nitroglycerin resulting in improved exercise tolerance, or peripherally limited, defined as no improvement in exercise tolerance despite reduction in pulmonary capillary wedge pressure after sublingual nitroglycerin. After baseline testing, subjects will be randomized to either whole body cycle exercise supplemented with sublingual nitroglycerin to improve training responsiveness or isolated single leg exercise training for 4 months. After 4 months, subjects will repeat maximal exercise testing and invasive right heart catheterization to assess responses to 4 months of exercise training.

ELIGIBILITY:
Inclusion Criteria:

* signs and symptoms of heart failure
* an ejection fraction > 0.50
* objective evidence of diastolic dysfunction

Exclusion Criteria:

* age < 60 years
* BMI > 50 kg/m2
* PDE5 inhibitor use
* Severe valvular disease
* Severe COPD
* CKD 4 or higher
* Contra-indication to MRI.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Aerobic fitness | 4 months
  Change in peak VO2 after exercise training

SECONDARY OUTCOMES:
Cardiopulmonary hemodynamics | 4 months
  Change in exercise pulmonary capillary wedge pressure
Sympathetic activity | 4 months
  Change in muscle sympathetic activity
Leg blood flow | 4 months
  Change in leg blood flow assessed by Doppler velocities in femoral artery
Cardiac fibrosis | 4 months
  Change in T1 mapping times by cardiac MRI

CONTACTS AND LOCATIONS:
Locations (1):
- The Institute for Exercise and Environmental Medicine, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Babb TG, Balmain BN, Tomlinson AR, Hynan LS, Levine BD, MacNamara JP, Sarma S. Ventilatory limitation to exercise in patients with HFpEF and obesity: No room to breathe. Respir Physiol Neurobiol. 2026 Jan 27;341:104546. doi: 10.1016/j.resp.2026.104546. Online ahead of print. PMID 41615840
- [Derived] Babb TG, Balmain BN, Tomlinson AR, Hynan LS, Levine BD, MacNamara JP, Sarma S. Ventilatory Limitation to Exercise in Patients with HFpEF and Obesity: No room to breatheVentilatory Limited Exercise in HFpEF. Respir Physiol Neurobiol. 2026 Jan 27:104546. doi: 10.1016/j.resp.2026.104546. Online ahead of print. PMID 41610904
- [Derived] Leahy MG, Wakeham DJ, MacNamara JP, Brazile T, Abulimiti A, Hearon CM Jr, Samels M, Tomlinson AR, Balmain BN, Babb TG, Levine BD, Sarma S. Heart-Lung Interactions in HFpEF: Dynamic Hyperinflation and Exercise PCWP. JACC Heart Fail. 2025 Aug;13(8):102523. doi: 10.1016/j.jchf.2025.102523. Epub 2025 Jun 26. PMID 40578265
- [Derived] Skow RJ, Sarma S, MacNamara JP, Bartlett MF, Wakeham DJ, Martin ZT, Samels M, Nandadeva D, Brazile TL, Ren J, Fu Q, Babb TG, Balmain BN, Nelson MD, Hynan LS, Levine BD, Fadel PJ, Haykowsky MJ, Hearon CM Jr. Identifying the Mechanisms of a Peripherally Limited Exercise Phenotype in Patients With Heart Failure With Preserved Ejection Fraction. Circ Heart Fail. 2024 Aug;17(8):e011693. doi: 10.1161/CIRCHEARTFAILURE.123.011693. Epub 2024 Jul 25. PMID 39051098
- [Derived] Sarma S, MacNamara JP, Balmain BN, Hearon CM Jr, Wakeham DJ, Tomlinson AR, Hynan LS, Babb TG, Levine BD. Challenging the Hemodynamic Hypothesis in Heart Failure With Preserved Ejection Fraction: Is Exercise Capacity Limited by Elevated Pulmonary Capillary Wedge Pressure? Circulation. 2023 Jan 31;147(5):378-387. doi: 10.1161/CIRCULATIONAHA.122.061828. Epub 2022 Dec 16. PMID 36524474